CLINICAL TRIAL: NCT06109545
Title: Validation of Doppler Ultrasound, CT Parameters Versus Laparoscopic Scoring in Assessment of Suspicious Ovarian Malignancy
Brief Title: Doppler Ultrasound and CT Versus Laparoscopy in Assessment of Ovarian Malignancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: SM.MD
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer, Doppler, CT, Laparoscopy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with suspicion of ovarian malignancy: Women with suspicion of ovarian malignancy depending on ultrasound, CT, MRI and CA 125
  Interventions: Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Laparoscopy — Patients included in this study will have diagnostic laparoscopy type WOLF done after checking all above ultrasound parameters of malignant tumor. This procedure will be done under general anathesia then a verses needle will be used at umbilicus or at palmer point if the mass is large or in cases of umbilical hernia or previous abdominal or pelvic surgery, then Fagotti criteria will be assessed
  Other Names: Laparoscopic Fagotti scoring

SUMMARY:
The aim of this study is to assess validation of ultrasound (± Doppler) parameters in the diagnosis of suspicious ovarian malignant tumors and laparoscopic assessment of these findings according to Fagotti score evaluation of suspicious malignant tumors

DETAILED DESCRIPTION:
The aim of this study is to asses validation of ultrasound (± Doppler) parameters in the diagnosis of suspicious ovarian malignant tumors and laparoscopic assessment of these findings according to Fagotti score evaluation of suspicious malignant tumors

ELIGIBILITY:
Inclusion Criteria:

1. all patients with clinical or radiological suspicion of ovarian cancer.
2. at least one of clinical presentation of suspected or advanced ovarian cancer and performed ultrasound or CT or MRI that detect a pelvic mass and CA125 is more than 200 UL/ML.
3. patients with eastern Cooperative Oncology Group status from 0 to 3.

Exclusion Criteria:

1. the women outside the age group in our study.
2. any known malignancy at other sites.
3. uncompliant patients who have severed uncontrolled infection or any other medical problem.
4. any previous major surgery.
5. patients who refuse to give an informed consent to do laparoscopy.
6. pregnancy and its complications.

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women with suspicious ovarian malignancy
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2023-06-24 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Fagotti score | Al time of laparoscopy
  Laparoscopic staging of suspicious ovarian mass

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Madany, MSc, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided